CLINICAL TRIAL: NCT05271175
Title: Accelerated Intermittent Theta Burst Stimulation in Smoking Cessation: A Randomized Controlled Study
Brief Title: Accelerated iTBS in Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus rTMS Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08.2019CY
Record Dates: First submitted 2022-02-04; First posted 2022-03-08 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Nicotine Dependence; Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Active TMS & Neutral videos (Experimental): Received active iTBS stimulation while watching neutral videos
  Interventions: Device: Active intermittent theta burst stimulation
- Active TMS & Smoking videos (Experimental): Received active iTBS stimulation while watching smoking-related videos
  Interventions: Device: Active intermittent theta burst stimulation
- Sham TMS & Smoking videos (Sham Comparator): Received sham stimulation while watching smoking-related videos
  Interventions: Device: Sham intermittent theta burst stimulation

INTERVENTIONS:
Device: Active intermittent theta burst stimulation — An accelerated iTBS (aiTBS) treatment (4 sessions with 30 minutes break between them) was administered daily for a 5-day period over the left DLPFC using the MagVenture Cool-B65 Active/Placebo (A/P) coil.
  Arms: Active TMS & Neutral videos; Active TMS & Smoking videos
Device: Sham intermittent theta burst stimulation — An accelerated iTBS (aiTBS) treatment (4 sessions with 30 minutes break between them) was administered daily for a 5-day period over the left DLPFC using the MagVenture Cool-B65 Active/Placebo (A/P) coil. The MagVenture Cool-B65 Active/Placebo (A/P) coil is designed to support true "double blinded" clinical trials as it can produce active and placebo stimulation by flipping the coil and can mimic tapping sensation during placebo condition During the sham condition, the coil produced the same sound as the real active condition but did not deliver any stimulation on the side of the participant's skull.
  Arms: Sham TMS & Smoking videos

SUMMARY:
Cigarette smoking is one of the foremost causes of preventable disease and premature death. In 2014, 68% of adult smokers wanted to quit smoking and in 2017, 55.1% of adult smokers had made a quit attempt. However, only a small percentage of adult smokers (7,4%) achieved to quit smoking.

Transcranial magnetic stimulation (TMS) is a novel, powerful, non-invasive brain stimulation therapy. This study used Theta Burst Stimulation (TBS), a newer form of rTMS protocol that can be delivered in a shorter duration compared to the standard rTMS protocol, while delivering a comparable number of pulses. It is a tolerable, powerful, and useful tool in non-invasive brain stimulation therapies.

This double-blind randomized control trial evaluated the efficacy of 4 iTBS sessions per day during 5 consecutive days over the left DLPFC in smoking cessation. Moreover, it investigated whether the exposure to smoking-related cues during the rTMS treatment, compared to neutral cues impact cigarette craving.

DETAILED DESCRIPTION:
Cigarette smoking is one of the foremost causes of preventable disease and premature death. In 2014, 68% of adult smokers wanted to quit smoking and in 2017, 55.1% of adult smokers had made a quit attempt. However, only a small percentage of adult smokers (7,4%) achieved to quit smoking. Behavioral and psychological interventions, pharmacological interventions as well as nicotine replacement therapy are some of the most used interventions for smoking cessation with medium to low success rates. Nonetheless, in recent years there has been growing interest in new, alternative, and effective treatments for smoking cessation.

Transcranial magnetic stimulation (TMS) is a novel, powerful, non-invasive brain stimulation therapy. TMS non-invasively (transcranially) delivers magnetic pulses to a brain region, inducing electric a current that can depolarize neurons and induce action potentials. This study used Theta Burst Stimulation (TBS), a newer form of rTMS protocol that can be delivered in a shorter duration compared to the standard rTMS protocol, while delivering a comparable number of pulses. It is a tolerable, powerful, and useful tool in non-invasive brain stimulation therapies.

This double-blind randomized control trial evaluated the efficacy of 4 iTBS sessions per day during 5 consecutive days over the left DLPFC in smoking cessation. Moreover, it investigated whether the exposure to smoking-related cues during the rTMS treatment, compared to neutral cues impact cigarette craving. The investigators hypothesized that twenty sessions of accelerated theta burst simulation over the left DLPFC while exposed to smoking-related cues, would reduce cigarette consumption and cigarette cravings, accompanied by reduced stress and motivation to quit smoking, compared to both active and sham stimulation with neutral-cues.

A total of 104 cigarettes smokers, who wanted to quit smoking, were enrolled and were randomly divided into the three experimental groups: the first group received active aiTBS stimulation while watching neutral videos, the second group received active aiTBS stimulation while watching smoking-related videos and the last group received sham stimulation while watching smoking-related videos. Primary and secondary measurements were performed at the baseline, during the treatment period, at one week, one month and six months post rTMS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-70
2. native or fluent Greek speaker.

Exclusion Criteria:

1. mental objects or implants in the brain, skull or near head (e.g., pacemakers, metal plates)
2. past or current of diagnosis of neurological or psychiatric disorder
3. use of psychiatric medication
4. past or current drug or alcohol abuse, other than nicotine
5. use of IQOS ("I Quit Original Smoking") or electronic cigarettes (e-cigarettes).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sack, Principal Investigator — Maastricht University, The Netherlands
Locations (1):
- Cyprus rTMS, Larnaca, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mikellides G, Michael P, Psalta L, Stefani A, Schuhmann T, Sack AT. Accelerated Intermittent Theta Burst Stimulation in Smoking Cessation: Placebo Effects Equal to Active Stimulation When Using Advanced Placebo Coil Technology. Front Psychiatry. 2022 May 24;13:892075. doi: 10.3389/fpsyt.2022.892075. eCollection 2022. PMID 35686190

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Started | 34 | 33 | 37
Completed | 29 | 30 | 30
Not Completed | 5 | 3 | 7
Period: One Week Follow up
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Started | 29 | 30 | 30
Completed | 19 | 23 | 25
Not Completed | 10 | 7 | 5
Not completed — Lost to Follow-up | 10 | 7 | 5
Period: One Month Follow up
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Started (Αll participants who completed the study (n=89) were asked to complete the one-month follow-up, regardless of whether they completed the one-week follow-up.) | 29 | 30 | 30
Completed | 17 | 23 | 21
Not Completed | 12 | 7 | 9
Not completed — Lost to Follow-up | 12 | 7 | 9
Period: Six Months Follow up
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Started (Αll participants who completed the study (n=89) were asked to complete the six-months follow-up, regardless of whether they completed the one-month follow-up.) | 29 | 30 | 30
Completed | 21 | 28 | 28
Not Completed | 8 | 2 | 2
Not completed — Lost to Follow-up | 8 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos | Total
Number analyzed (Participants) | 29 | 30 | 30 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.52 (13.05) | 42.93 (14.42) | 47.43 (12.72) | 45.62 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 12 | 29
  Male | 22 | 20 | 18 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Education [Mean (Standard Deviation); unit: years] | 14.07 (3.95) | 14.43 (3.77) | 13.60 (3.27) | 14.03 (3.65)
Occupation [Count of Participants; unit: Participants]
  Private employee | 13 | 19 | 22 | 54
  Public employee | 7 | 4 | 1 | 12
  Self-employed / freelancer | 5 | 1 | 4 | 10
  Unemployed | 2 | 1 | 0 | 3
  Retired | 2 | 4 | 3 | 9
  Student | 0 | 1 | 0 | 1
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes/day] | 27.55 (15.37) | 26.83 (12.86) | 30.00 (13.38) | 28.13 (13.80)
Types of cigarettes [Count of Participants; unit: Participants]
  Normal | 16 | 25 | 24 | 65
  Hand-rolled | 10 | 5 | 5 | 20
  Cigarillos | 1 | 0 | 0 | 1
  Mixed | 2 | 0 | 1 | 3
Years of smoking [Mean (Standard Deviation); unit: years] | 23.18 (9.82) | 23.13 (13.58) | 28.73 (12.21) | 25.06 (12.17)
If ever quitted [Count of Participants; unit: Participants]
  No | 9 | 10 | 11 | 30
  Yes | 20 | 20 | 19 | 59
How many times quitted [Mean (Standard Deviation); unit: quit attempts] | 0.90 (0.77) | 1.00 (1.11) | 1.20 (1.56) | 1.03 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Nicotine Consumption
Description: Τhe number of cigarettes participants usually smoke before the treatment.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: cigarettes/day
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
cigarettes/day | 27.55 (15.37) | 26.83 (12.86) | 30.00 (13.38)

2. Primary Outcome: Self-reported Nicotine Consumption
Description: Participants were required to record the number of cigarettes smoked after the completion of the 1st day of treatment until before the first session on the second day of treatment. Participants were asked not to smoke during the breaks of the 4 daily rTMS sessions
Time Frame: After 1st treatment day
Population: Two participants from the "Active TMS & Neutral videos" group and three participants from the "Active TMS & Smoking videos" group were outliers and were therefore excluded from the analyses.
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 27 | 27 | 30
cigarettes/day | 8.72 (8.97) | 8.67 (8.56) | 10.60 (7.49)

3. Primary Outcome: Self-reported Nicotine Consumption
Description: Participants were required to record the number of cigarettes smoked after the completion of the 2nd day of treatment until before the first session on the 3rd day of treatment. Participants were asked not to smoke during the breaks of the 4 daily rTMS sessions
Time Frame: After 2nd treatment day
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 27 | 29 | 30
cigarettes/day | 7.94 (8.13) | 7.07 (6.43) | 9.38 (7.90)

4. Primary Outcome: Self-reported Nicotine Consumption
Description: Participants were required to record the number of cigarettes smoked after the completion of the 3rd day of treatment until before the first session on the 4th day of treatment. Participants were asked not to smoke during the breaks of the 4 daily rTMS sessions
Time Frame: After 3rd treatment day
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 26 | 26 | 30
cigarettes/day | 5.92 (6.68) | 7.79 (8.61) | 8.20 (7.80)

5. Primary Outcome: Self-reported Nicotine Consumption
Description: Participants were required to record the number of cigarettes smoked after the completion of the 4th day of treatment until before the first session on the 5th day of treatment . Participants were asked not to smoke during the breaks of the 4 daily rTMS sessions
Time Frame: After 4th treatment day
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 26 | 27 | 30
cigarettes/day | 5.27 (7.51) | 4.67 (6.50) | 6.27 (7.84)

6. Primary Outcome: Carbon Monoxide (CO)- Evaluated Nicotine Consumption
Description: CO level was measured using the piCO Smokerlyzer breath carbon monoxide meter device prior to the first rTMS session.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 28 | 29 | 30
ppm | 23.64 (14.68) | 17.24 (10.17) | 21.13 (9.63)

7. Primary Outcome: Carbon Monoxide (CO)- Evaluated Nicotine Consumption
Description: The average of the four CO-levels, measured before each of the four sessions on Day 1.
Time Frame: Day 1
Measure: Mean (Standard Error); unit: ppm
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
ppm | 19.09 (12.14) | 14.83 (8.47) | 17.77 (7.88)

8. Primary Outcome: Carbon Monoxide (CO)- Evaluated Nicotine Consumption
Description: The average of the four CO-levels, measured before each of the four sessions on Day 2.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
ppm | 11.09 (9.69) | 9.94 (8.17) | 11.03 (7.50)

9. Primary Outcome: Carbon Monoxide (CO)- Evaluated Nicotine Consumption
Description: The average of the four CO-levels, measured before each of the four sessions on Day 3.
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
ppm | 9.98 (10.15) | 9.61 (6.63) | 8.85 (6.58)

10. Primary Outcome: Carbon Monoxide (CO)- Evaluated Nicotine Consumption
Description: The average of the four CO-levels, measured before each of the four sessions on Day 4.
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
ppm | 8.35 (8.44) | 8.58 (6.65) | 8.89 (6.96)

11. Primary Outcome: Carbon Monoxide (CO)- Evaluated Nicotine Consumption
Description: The average of the four CO-levels, measured before each of the four sessions on Day 5.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
ppm | 8.98 (9.68) | 8.03 (7.27) | 8.18 (7.02)

12. Primary Outcome: Nicotine Dependence
Description: Fagerström test for Nicotine Dependence (FTND) is a short, self-report measure that assesses nicotine dependence. It contains six questions, and the total score is calculated as a sum of these six questions. The scores vary from 0 to 10, with lower scores indicating lower dependence on nicotine.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 5.86 (2.26) | 6.03 (2.37) | 6.77 (2.27)

13. Primary Outcome: Nicotine Dependence
Description: as for outcome 12
Time Frame: End of the treatment (On the fifth day, after completing 20 TMS sessions)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 2.31 (2.62) | 2.03 (2.08) | 2.57 (2.69)

14. Primary Outcome: Nicotine Dependence
Description: as for outcome 12
Time Frame: 1 week follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 19 | 23 | 25
score on a scale | 1.79 (1.55) | 2.04 (2.49) | 2.64 (2.41)

15. Primary Outcome: Nicotine Dependence
Description: as for outcome 12
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 17 | 23 | 21
score on a scale | 3.35 (1.97) | 2.78 (2.80) | 3.38 (2.84)

16. Primary Outcome: Nicotine Dependence
Description: as for outcome 12
Time Frame: 6 months follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 21 | 28 | 28
score on a scale | 3.71 (2.43) | 3.32 (2.74) | 3.96 (2.57)

17. Primary Outcome: Momentary Craving
Description: The Visual Analogue Scale (VAS) is a psychometric measurement instrument that measures symptom severity on a continuous scale. The VAS can be quickly and repeatedly administered between tasks and it has been used extensively in smoking research with TMS. We used the VAS to assess smoking craving by asking participants to respond to the question "How much do you want to smoke right now?", on a scale from 0 "no craving" to 100 "most craving ever experienced" by choosing a response on a visual scale given in front of them on a tablet.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 24.21 (30.64) | 30.87 (28.63) | 25.70 (30.42)

18. Primary Outcome: Momentary Craving
Description: The Visual Analogue Scale (VAS) is a psychometric measurement instrument that measures symptom severity on a continuous scale. The VAS can be quickly and repeatedly administered between tasks and it has been used extensively in smoking research with TMS. We used the VAS to assess smoking craving by asking participants to respond to the question "How much do you want to smoke right now?", on a scale from 0 "no craving" to 100 "most craving ever experienced" by choosing a response on a visual scale given in front of them on a tablet.
  The average of the eight VAS scores, measured prior and post each of the four sessions on Day 1.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 24.55 (20.66) | 33.13 (22.12) | 29.03 (28.59)

19. Primary Outcome: Momentary Craving
Description: The Visual Analogue Scale (VAS) is a psychometric measurement instrument that measures symptom severity on a continuous scale. The VAS can be quickly and repeatedly administered between tasks and it has been used extensively in smoking research with TMS. We used the VAS to assess smoking craving by asking participants to respond to the question "How much do you want to smoke right now?", on a scale from 0 "no craving" to 100 "most craving ever experienced" by choosing a response on a visual scale given in front of them on a tablet.
  The average of the eight VAS scores, measured prior and post each of the four sessions on Day 2.
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 15.62 (16.69) | 23.54 (18.88) | 21.87 (24.12)

20. Primary Outcome: Momentary Craving
Description: The Visual Analogue Scale (VAS) is a psychometric measurement instrument that measures symptom severity on a continuous scale. The VAS can be quickly and repeatedly administered between tasks and it has been used extensively in smoking research with TMS. We used the VAS to assess smoking craving by asking participants to respond to the question "How much do you want to smoke right now?", on a scale from 0 "no craving" to 100 "most craving ever experienced" by choosing a response on a visual scale given in front of them on a tablet.
  The average of the eight VAS scores, measured prior and post each of the four sessions on Day 3.
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 12.45 (15.33) | 22.32 (19.87) | 17.48 (21.78)

21. Primary Outcome: Momentary Craving
Description: The Visual Analogue Scale (VAS) is a psychometric measurement instrument that measures symptom severity on a continuous scale. The VAS can be quickly and repeatedly administered between tasks and it has been used extensively in smoking research with TMS. We used the VAS to assess smoking craving by asking participants to respond to the question "How much do you want to smoke right now?", on a scale from 0 "no craving" to 100 "most craving ever experienced" by choosing a response on a visual scale given in front of them on a tablet.
  The average of the eight VAS scores, measured prior and post each of the four sessions on Day 4.
Time Frame: Day 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 9.16 (13.12) | 20.14 (18.41) | 14.44 (19.18)

22. Primary Outcome: Momentary Craving
Description: The Visual Analogue Scale (VAS) is a psychometric measurement instrument that measures symptom severity on a continuous scale. The VAS can be quickly and repeatedly administered between tasks and it has been used extensively in smoking research with TMS. We used the VAS to assess smoking craving by asking participants to respond to the question "How much do you want to smoke right now?", on a scale from 0 "no craving" to 100 "most craving ever experienced" by choosing a response on a visual scale given in front of them on a tablet.
  The average of the eight VAS scores, measured prior and post each of the four sessions on Day 5.
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 10.57 (15.74) | 16.08 (16.14) | 10.46 (13.13)

23. Primary Outcome: General Craving
Description: Tobacco Craving Questionnaire-Short Form (TCQ-SF) is a self-report measure that assesses tobacco craving in four dimensions. Each factor scale contains three items. TCQ-SF items were rated on a Likert scale of 1 (strongly disagree) to 7 (strongly agree). Total scores vary from 12 to 84, by summing the 12 items and the scores for each factor scale vary from 3 to 21 by summing the three items in each factor scale. A high score indicates high tobacco craving.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
Total score | 45.38 (17.95) | 52.03 (16.20) | 43.83 (17.25)

24. Primary Outcome: General Craving
Description: as for outcome 23
Time Frame: End of the treatment (On the fifth day, after completing 20 TMS sessions)
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
Total score | 30.93 (17.05) | 31.97 (14.61) | 28.63 (13.10)

25. Primary Outcome: General Craving
Description: as for outcome 23
Time Frame: 1 week follow up
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 19 | 23 | 25
Total score | 29.84 (14.18) | 32.17 (21.57) | 27.28 (14.82)

26. Primary Outcome: General Craving
Description: as for outcome 23
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 17 | 23 | 21
Total score | 37.06 (17.94) | 30.61 (19.63) | 35.24 (20.63)

27. Primary Outcome: General Craving
Description: as for outcome 23
Time Frame: 6 months follow up
Measure: Mean (Standard Deviation); unit: Total score
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 21 | 28 | 28
Total score | 51.52 (19.50) | 38.32 (18.22) | 44.68 (22.34)

28. Secondary Outcome: Perceived Stress
Description: Perceived Stress Scale-4 (PSS-4) is a self-report measure that is used to assess psychological stress. PSS-4 items were rated on a Likert scale, ranging from 0 to 4, with those on the positive subscale scored in reverse and the total score was calculated as a sum of these items. The scores vary from 0-16, with a higher score indicating higher perceived stress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 5.97 (2.18) | 6.53 (2.40) | 5.60 (1.98)

29. Secondary Outcome: Perceived Stress
Description: as for outcome 28
Time Frame: End of the treatment (On the fifth day, after completing 20 TMS sessions)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 29 | 30 | 30
score on a scale | 5.21 (2.47) | 5.90 (2.34) | 4.60 (1.96)

30. Secondary Outcome: Perceived Stress
Description: as for outcome 28
Time Frame: 1 week follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 19 | 23 | 25
score on a scale | 4.42 (2.59) | 6.00 (2.66) | 4.76 (2.35)

31. Secondary Outcome: Perceived Stress
Description: as for outcome 28
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 17 | 23 | 21
score on a scale | 4.06 (2.66) | 5.57 (2.13) | 3.52 (2.48)

32. Secondary Outcome: Perceived Stress
Description: as for outcome 28
Time Frame: 6 months follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 21 | 28 | 28
score on a scale | 4.67 (1.88) | 5.75 (2.05) | 4.75 (2.52)

33. Secondary Outcome: Motivation to Quit Smoking
Description: Participants were asked to estimate how motivated they were to quit smoking from 0% to 100%. Τhe possible answers were: 0%, 25%, 50%, 75% and 100%. Higher values reflect greater motivation to quit smoking.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 27 | 27 | 30
score on a scale | 77.78 (21.18) | 82.41 (18.10) | 80.83 (20.43)

34. Secondary Outcome: Motivation to Quit Smoking
Description: as for outcome 33
Time Frame: End of the treatment (On the fifth day, after completing 20 TMS sessions)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 27 | 27 | 30
score on a scale | 82.41 (20.59) | 84.26 (19.79) | 80.83 (23.38)

35. Secondary Outcome: Motivation to Quit Smoking
Description: as for outcome 33
Time Frame: 1 week follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 19 | 23 | 25
score on a scale | 72.37 (23.41) | 77.17 (30.07) | 75.00 (27.95)

36. Secondary Outcome: Motivation to Quit Smoking
Description: as for outcome 33
Time Frame: 1 month follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 17 | 23 | 21
score on a scale | 47.06 (31.72) | 70.65 (37.43) | 52.38 (38.65)

37. Secondary Outcome: Motivation to Quit Smoking
Description: as for outcome 33
Time Frame: 6 months follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
Number analyzed (Participants) | 21 | 28 | 28
score on a scale | 41.67 (34.76) | 67.86 (32.53) | 52.68 (34.92)

ADVERSE EVENTS:
Time Frame: 1 week
Description: Participants were asked to daily report (during the 5-day treatment period) the adverse events they may have had experienced.
Arm/Group | Active TMS & Neutral Videos | Active TMS & Smoking Videos | Sham TMS & Smoking Videos
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 11/29 | 5/30 | 7/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active TMS & Neutral Videos (N=29) | Active TMS & Smoking Videos (N=30) | Sham TMS & Smoking Videos (N=30)
Mild headache (General disorders) | 2 (2) | 4 (4) | 1 (1)
Sleepiness (General disorders) | 3 (3) | 0 (0) | 2 (2)
Insomnia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (General disorders) | 0 (0) | 0 (0) | 1 (1)
Numbness on stimulation site (General disorders) | 1 (1) | 0 (0) | 0 (0)
Tension (General disorders) | 1 (1) | 0 (0) | 1 (1)
Lightheadedness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Coghiness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Numbness on stimulation site & Forgetfulness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Numbness on stimulation site & Sleepiness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mild headache & Sleepiness (General disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT05271175/Prot_SAP_001.pdf